CLINICAL TRIAL: NCT00296244
Title: Steroid Free Immunosuppression in Liver Transplantation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: CERL080AUS29
Record Dates: First submitted 2006-02-23; First posted 2006-02-24 (Estimated); Results first posted 2012-11-19 (Estimated); Last update posted 2012-11-19 (Estimated); Status verified 2012-10

CONDITIONS: Liver Cirrhosis; Liver Transplant Disorder
Keywords: steroid-free immunosuppression; liver transplantation
MeSH Terms: conditions — Liver Cirrhosis | interventions — Steroids; Methylprednisolone; Methylprednisolone Hemisuccinate; Prednisone; Basiliximab; Tacrolimus; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Steroid -free immunosuppression (Other): Study group - Basiliximab, Tacrolimus, Enteric-coated Mycophenolic acid (EC-MPA)
  Interventions: Drug: Basiliximab; Drug: Tacrolimus; Drug: Enteric-coated Mycophenolic acid (EC-MPA)
- Steroid containing immunosuppression (Other): Control group- Basiliximab, Tacrolimus, EC-MPA, steroids
  Interventions: Drug: Steroids; Drug: Basiliximab; Drug: Tacrolimus; Drug: Enteric-coated Mycophenolic acid (EC-MPA)

INTERVENTIONS:
Drug: Steroids — Patients randomized to Control group shall be administered steroids as methylprednisolone (Solumedrol) 1000 mg IV during the anhepatic phase. Methylprednisolone will be continued according to the following taper schedule: 50 mg IV every 6 hrs on day 1; 40 mg IV every 6hrs on day 2; 30 mg IV every 6 hrs on day 3; 20 mg IV every 6 hrs on day 4; 20 mg IV every 12 hrs on day 5; and Prednisone 20 mg by mouth or Naso-gastric tube (NGT) on day 6. Prednisone shall be tapered slowly starting at 1 month post-OLT and weaned off completely by 6 months post-OLT.
  Other Names: Methylprednisolone (Solumedrol); Prednisone
  Arms: Steroid containing immunosuppression
Drug: Basiliximab — Basiliximab shall be given as induction therapy at 20 mg IV bolus intra-operatively and on the 4th day after transplantation.
  Other Names: Simulect
Drug: Tacrolimus — Tacrolimus shall be used as the main maintenance immuno-suppressive drug. It will be given at a dose of 0.15mg/ kg/ day by mouth or through a naso-gastric tube (NGT), starting not earlier than 24 after the transplant but within 48 hrs after reperfusion. The dose shall be adjusted to achieve a trough level of 10-15 ng/ml during the first 30 days after transplantation and lowered to 5-10 ng/ml, thereafter.
  Other Names: Prograf
Drug: Enteric-coated Mycophenolic acid (EC-MPA) — This drug may be given in combination with calcineurin inhibitors (tacrolimus) and steroids for maintenance immuno-prophylaxis to prevent rejection. They are particularly useful in recipients with renal dysfunction and neurotoxicity, when there is a need to reduce dose or delay introduction of calcineurin inhibitors. This drug is given at 720 mg PO BID for 3 months.
  Other Names: Myfortic

SUMMARY:
The purpose of this study is to determine whether steroid-related complications can be avoided by using steroid-free immuno-suppressive drug regimen after liver transplantation.

DETAILED DESCRIPTION:
Steroids have remained a standard part of post-transplant immunosuppression, both for prevention and treatment of rejection. However, steroids have been shown to cause long-term adverse effects, such as: susceptibility to infection, obesity, hypertension, hyperlipidemia, diabetes, osteopenia, cataracts and growth retardation in children. They have also been implicated in accelerating Hepatitis C virus (HCV) re-infection post-liver transplantation.

Several studies have shown that early steroid reduction or withdrawal could be done safely to alleviate many steroid-related adverse effects after liver transplantation (OLT).

This is a prospective controlled randomized trial on adult patients who will undergo primary OLT at Thomas Jefferson University Hospital (TJUH).

Forty consecutive OLT recipients shall be randomized into two groups.

* Control group- immuno-suppressive drug regimen consisting of basiliximab (Simulect), tacrolimus (Prograf), Mycophenolic acid (Myfortic), and steroids
* Study group- immuno-suppressive drug regimen consisting of basiliximab, tacrolimus, Mycophenolic acid (Myfortic) without steroids

Basiliximab will be given at 20 mg IV bolus intra-operatively and on the 4th day after transplantation. Tacrolimus shall be administered at a dose of 0.15mg/ kg/ day by mouth or through a naso-gastric tube (NGT), starting not earlier than 24 after the transplant but within 48 hrs after reperfusion. The dose shall be adjusted to achieve a trough level of 10-15 ng/ml during the first 30 days after transplantation and lowered to 5-10 ng/ml, thereafter. Patients randomized to the control group shall be administered methylprednisolone (Solumedrol) 1000 mg IV during the anhepatic phase. Methylprednisolone will be continued according to the following taper schedule: 50 mg IV every 6 hrs on day 1; 40 mg IV every 6hrs on day 2; 30 mg IV every 6 hrs on day 3; 20 mg IV every 6 hrs on day 4; 20 mg IV every 12 hrs on day 5; and Prednisone 20 mg by mouth or NGT on day 6. Prednisone shall be tapered slowly starting at 1 month post-OLT and weaned off completely by 6 months post-OLT. Enteric-coated mycophenolic acid or EC-MPA (Myfortic) will be added to the regimen, particularly in patients with renal impairment or neuro-toxicity to minimize the dose and effects of tacrolimus. It will be started at 720 mg P.O. 2x/ day immediately post-transplant and shall be given for a period of 3 months.

Primary end points of this study at 6 months post-transplant include: graft and patient survival rates, and incidence of acute rejection and therapy employed to treat rejection. Secondary end points include: adverse effects of steroids, particularly, diabetes, obesity, hyperlipidemia, and hypertension; incidence and severity of HCV recurrence, and incidence of infectious complications.

Blood samples of HCV recipients shall be collected on day of surgery, 2 weeks, 1 month, 3 months, and 6 months post-OLT as per TJUH Liver Transplant Protocol. Sera shall be stored at -80C and will be used for quantitative HCV RNA levels by quantitative polymerase chain reaction.

Protocol liver biopsy shall be performed at the time of surgery, between 7-21 days post-OLT and at approximately 3 months after transplantation or as clinically indicated by elevated liver function test results.

Acute rejection shall be treated initially by increasing the tacrolimus dose to achieve a level 15-20 ng/ml for 48 hrs. If liver function test results will not show improvement by the 3rd day after increasing tacrolimus dose, a biopsy should be performed. Only biopsy proven rejection shall be treated according to the following protocol. Mild to moderate rejection shall be treated in the study group with methylprednisolone 1 gm IV with tapering doses of steroid as described above. Steroids shall be discontinued after the completion of the taper. In the control group, methylprednisolone 1 gm IV shall be followed by tapering doses and by prednisone 20 mg once daily, which shall be progressively reduced accordingly. The protocol shall also include a repeat biopsy if there is no improvement in the liver function test at the end of steroid taper. Severe rejection or steroid resistant rejection shall be treated with OKT3 at 5mg IV/ day for 5-10 days after pre-medication.

Recipients with HCV recurrence shall be treated according to TJUH Liver Transplant protocol as follows. Abnormal liver function tests should be evaluated by hepatic imaging to exclude anatomic abnormality. If none, liver biopsy will be done. If liver biopsy shows > grade 4 (inflammation more than mild) or > stage 1 (fibrosis), consider antiviral treatment consisting of Peg-Interferon alpha-2a 180mcg subcutaneously weekly for two weeks. If patient tolerates peg-interferon from hematologic and neuro-psychiatric standpoint, continue peg-interferon, and add ribavirin. Refer to protocol for dosing. Total duration of therapy is 48 weeks.

Follow up period for primary analysis will be six (6) months.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients between 18 and 72 years of age
* Male or female patients who are primary cadaveric liver transplant recipients
* Cold ischemia time must be <20 hours
* Females capable of becoming pregnant must have a negative pregnancy test at baseline and are required to practice an approved method of birth control for the duration of the study and for a period of three months following discontinuation of study medication
* Patient has given written informed consent to participate in the study

Exclusion Criteria:

* Patients meeting any of the following criteria at baseline will be excluded from study participation
* Patients who have previously received an organ transplant
* Patients who are recipients of a multiple organ transplants
* Women of childbearing potential not using the contraception method(s) specified in this study, as well as women who are breastfeeding
* Known sensitivity to Simulect or class of Simulect
* Patients with severe medical condition(s) that in the view of the investigator prohibits participation in the study
* Use of any other investigational agent in the last 30 days

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-02; Primary Completion 2008-05 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Gerardo B Ramirez, M.D., Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between February 2006 and November 2007,at Thomas Jefferson University, 40 adult orthotopic liver transplantation recipients were enrolled in the study and 20 recipients were randomized in each group.
Pre-assignment Details: One recipient in the Steroid free group required re-transplantation and died within 1 month after the 2nd OLT, and was subsequently excluded from analysis.
Groups:
- Control Group: Control group- basiliximab (Simulect), tacrolimus (Prograf), EC-MPA (Myfortic)with steroids
- Study Group: Study group- basiliximab (Simulect), tacrolimus (Prograf), EC-MPA (Myfortic)
Period: Overall Study
Arm/Group | Control Group | Study Group
Started | 20 | 20
Completed | 20 | 19
Not Completed | 0 | 1
Not completed — Underwent retransplant | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Control Group: Control group -basiliximab, tacrolimus, EC-MPA, steroids
- Study Group: Study group- basiliximab, tacrolimus, EC-MPA
- Total: Total of all reporting groups
Arm/Group | Control Group | Study Group | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 18 | 37
  >=65 years | 1 | 2 | 3
Age Continuous [Mean (Standard Deviation); unit: years] | 50.40 (2.6) | 56.2 (1.1) | 53 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 15 | 15 | 30
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Graft Survival Rate
Description: Percentage of recipients whose liver grafts are still working at the end of 1 and 2 years.
Time Frame: 1 and 2 years
Measure: Number; unit: percentage of participants
Groups:
- Control Group: Control group-basiliximab, tacrolimus, EC-MPA, steroids
Arm/Group | Control Group | Study Group
Number analyzed (Participants) | 20 | 19
percentage of participants
  1-year graft survival rate | 100 | 94.7
  2-year graft survival rate | 90 | 84

2. Primary Outcome: Patient Survival Rate
Description: Percentage of recipients who are still alive at the end of 1 and 2 years.
Time Frame: 1 and 2 years
Measure: Number; unit: Percentage of participants
Arm/Group | Control Group | Study Group
Number analyzed (Participants) | 20 | 19
Percentage of participants
  1-year patient survival rate | 100 | 94.7
  2-year patient survival rate | 90 | 84

3. Primary Outcome: Acute Rejection Rate
Description: Biopsy proven acute rejection defined by biochemical and histological changes as well as the need for temporary steroid use occurred in 1 patient in each group both of which were steroid responsive
Time Frame: 6 months post-transplant
Measure: Number; unit: Percentage of participants
Groups:
- Study Group: Study group -basiliximab, tacrolimus, EC-MPA
Arm/Group | Control Group | Study Group
Number analyzed (Participants) | 20 | 19
Percentage of participants | 5 | 5

4. Secondary Outcome: Infection as an Adverse Effect of Steroids
Description: Incidence of bacterial infection was similar in the control group as well as study group, 4 patients in both groups had infection
Time Frame: 3 months post-transplant
Measure: Number; unit: Percentage of participants
Groups:
- Control Group: Control group)-basiliximab, tacrolimus, EC-MPA, steroids
Arm/Group | Control Group | Study Group
Number analyzed (Participants) | 20 | 19
Percentage of participants | 20 | 21

5. Secondary Outcome: Incidence and Severity of HCV Recurrence Post-OLT
Description: The incidence and severity of HCV recurrence based on Hepatitis C PCR levels and protocol liver biopsy findings were found to be similar between the 2 groups.
Time Frame: 6 months post-transplant
Population: Only patients with HCV cirrhosis as the main indication for OLT were included in this analysis
Measure: Number; unit: Percentage of participants
Arm/Group | Control Group | Study Group
Number analyzed (Participants) | 11 | 14
Percentage of participants | 27 | 29

6. Secondary Outcome: New-onset Diabetes Mellitus (NODM) as Secondary Outcome
Description: The incidence of new-onset Diabetes mellitus (NODM, based on percentage of previously non-diabetic patients who developed DM post-transplantation, was similar between the 2 groups.
Time Frame: 6 months
Measure: Number; unit: Percentage of participants
Groups:
- Control Group: Control group- basiliximab, tacrolimus, EC-MPA, steroids
- Study Group: Study group - basiliximab, tacrolimus, EC-MPA
Arm/Group | Control Group | Study Group
Number analyzed (Participants) | 20 | 19
Percentage of participants | 40 | 42

ADVERSE EVENTS:
Time Frame: Adverse data were collected at 1 and 2 years follow-up.
Arm/Group | Control Group | Study Group
Serious Adverse Events (participants affected / at risk) | 2/20 | 3/19
Other Adverse Events (participants affected / at risk) | 16/20 | 17/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Group (N=20) | Study Group (N=19)
Death (General disorders) | 2 (2) | 3 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Control Group (N=20) | Study Group (N=19)
Acute rejection (Immune system disorders) | 1 (1) | 1 (1)
Infection (Infections and infestations) | 4 (4) | 4 (4)
New-onset Diabetes Mellitus (NODM) (Endocrine disorders) | 8 (8) | 8 (8)
Hepatitis C Recurrence (Hepatobiliary disorders) | 3/11 (3) | 4/14 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes